CLINICAL TRIAL: NCT00921518
Title: Prevention of Acute Kidney Injury in Cardiac Surgery Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Community Medical Center, Scranton, PA (Other)
Responsible Party: Principal Investigator, Judith L. Kristeller, Associate Professor, Community Medical Center, Scranton, PA
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CMC AKICS
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-03

CONDITIONS: Kidney Injury
Keywords: Cardiac surgery; Sodium bicarbonate; Acute kidney injury; Saline
MeSH Terms: conditions — Acute Kidney Injury | interventions — Sodium Chloride; Saline Solution; Sodium Bicarbonate; Bicarbonates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Saline (Placebo Comparator): This group will receive isotonic saline at 3 ml/kg/hr for one hour pre-operatively until the patient is started on cardiopulmonary bypass. Then the infusion will be reduced to 1 ml/kg/hr throughout cardiopulmonary bypass and for six hours following cardiopulmonary bypass.
  Interventions: Drug: 0.9% Sodium Chloride (Placebo)
- Sodium Bicarbonate (Active Comparator): This arm two will receive sodium bicarbonate 150mEq in 850ml of a 5% dextrose solution at 3 ml/kg/hr for one hour pre-operatively until the patient is started on cardiopulmonary bypass. Then the infusion will be reduced to 1 ml/kg/hr throughout cardiopulmonary bypass and for six hours following cardiopulmonary bypass.
  Interventions: Drug: Sodium Bicarbonate

INTERVENTIONS:
Drug: 0.9% Sodium Chloride (Placebo) — 0.9% Sodium Chloride (placebo) will infuse at 3 ml/kg/hr for one hour pre-operatively until the patient is started on cardiopulmonary bypass. Then the infusion will be reduced to 1 ml/kg/hr throughout cardiopulmonary bypass and for six hours following cardiopulmonary bypass.
  Other Names: Normal Saline
  Arms: Normal Saline
Drug: Sodium Bicarbonate — Group two will receive sodium bicarbonate 150mEq in 850ml of a 5% dextrose solution at 3 ml/kg/hr for one hour pre-operatively until the patient is started on cardiopulmonary bypass. Then the infusion will be reduced to 1 ml/kg/hr throughout cardiopulmonary bypass and for six hours following cardiopulmonary bypass.
  Other Names: Bicarbonate
  Arms: Sodium Bicarbonate

SUMMARY:
Acute kidney injury (AKI) has no uniform criteria, but is commonly defined as an increase in serum creatinine concentration by at least 25% from baseline. It occurs in 30% of patients following cardiac surgery, and at least 50% of patients with underlying renal insufficiency. Patients who have a reduced creatinine clearance pre-operatively are at the greatest risk of developing post-operative AKI. The purpose of the current study is to determine if intravenous hydration with either isotonic saline or sodium bicarbonate 150 mEq/L is effective at preventing post-operative AKI in patients with baseline kidney insufficiency and who are undergoing cardiac surgery using cardiopulmonary bypass. The study hypothesis is that an infusion of sodium bicarbonate 150 mEq/L will be more effective than isotonic saline in reducing the incidence of post-operative AKI in cardiac surgery patients with a preoperative glomerular filtration rate (GFR) less than 60 ml/min/1.73m2.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, prospective, double-blinded. The study will take place at Community Medical Center in Scranton, Pennsylvania. The inclusion criteria are patients undergoing elective, urgent, or emergent cardiac surgery using cardiopulmonary bypass and having a baseline GFR less than 60 ml/min/1.73m2 estimated using the Modification of Diet in Renal Disease equation. Patients will be excluded from the study if they have cardiogenic shock (defined as a cardiac index less 2 L/min/m2 despite high dose inotropes or the need for intra-aortic balloon pump), end-stage kidney disease requiring dialysis, received an infusion of sodium bicarbonate on the same day as cardiac surgery, or if they are enrolled in a separate clinical research trial. This trial will involve two treatment groups. Group one will receive isotonic saline at 3 ml/kg/hr for one hour pre-operatively until the patient is started on cardiopulmonary bypass. Then the infusion will be reduced to 1 ml/kg/hr throughout cardiopulmonary bypass and for six hours following cardiopulmonary bypass. Group two will receive sodium bicarbonate 150mEq in 850ml of a 5% dextrose solution using the same infusion regimen as described above for isotonic saline. The primary efficacy outcome of the study will be the incidence of AKI postoperatively. Acute kidney injury will be defined as an increase in serum creatinine concentration by at least 25% from baseline or an absolute increase of 0.5 mg/dL at any time within the first five postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* elective, urgent, or emergent cardiac surgery using cardiopulmonary bypass
* baseline GFR less than 60 ml/min/1.73m2 estimated using the Modification of Diet in Renal Disease equation

Exclusion Criteria:

* cardiogenic shock (defined as a cardiac index less 2 L/min/m2 despite high dose inotropes or the need for intra-aortic balloon pump)
* end-stage kidney disease requiring dialysis
* received an infusion of sodium bicarbonate on the same day as cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith L Kristeller, PharmD, Principal Investigator — Wilkes University
Locations (1):
- Community Medical Center, Scranton, Pennsylvania, United States

REFERENCES:
- [Result] Kristeller JL, Zavorsky GS, Prior JE, Keating DA, Brady MA, Romaldini TA, Hickman TL, Stahl RF. Lack of effectiveness of sodium bicarbonate in preventing kidney injury in patients undergoing cardiac surgery: a randomized controlled trial. Pharmacotherapy. 2013 Jul;33(7):710-7. doi: 10.1002/phar.1262. Epub 2013 Apr 1. PMID 23553549

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Saline: This group will receive isotonic saline at 3 ml/kg/hr for one hour pre-operatively until the patient is started on cardiopulmonary bypass. Then the infusion will be reduced to 1 ml/kg/hr throughout cardiopulmonary bypass and for six hours following cardiopulmonary bypass.
  0.9% Sodium Chloride (Placebo): 3 ml/kg/hr for one hour pre-operatively until the patient is started on cardiopulmonary bypass. Then the infusion will be reduced to 1 ml/kg/hr throughout cardiopulmonary bypass and for six hours following cardiopulmonary bypass.
Period: Overall Study
Arm/Group | Normal Saline | Sodium Bicarbonate
Started | 48 | 44
Completed | 48 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Sodium Bicarbonate | Total
Number analyzed (Participants) | 48 | 44 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (11) | 72 (11) | 72 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 16 | 39
  Male | 25 | 28 | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Kidney Injury
Description: Acuge kidney injury is defined using the AKIN criteria
Time Frame: 5 days
Measure: Number; unit: participants
Arm/Group | Normal Saline | Sodium Bicarbonate
Number analyzed (Participants) | 48 | 44
participants | 20 | 14

ADVERSE EVENTS:
Arm/Group | Normal Saline | Sodium Bicarbonate
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/44
Other Adverse Events (participants affected / at risk) | 0/48 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Saline (N=48) | Sodium Bicarbonate (N=44)
Electrolyte Abnormalities (Endocrine disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes